CLINICAL TRIAL: NCT01827475
Title: Ibuprofen Versus Acetaminophen vs Their Combination in the Relief of Musculoskeletal Pain in the Emergency Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Professor and Vice Chair, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBNet119536
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: musculoskeletal pain; acetaminophen; ibuprofen
MeSH Terms: conditions — Pain; Musculoskeletal Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen (Active Comparator): Ibuprofen 800 mg
  Interventions: Drug: Ibuprofen
- Acetaminophen (Active Comparator): Acetaminophen 1 gm
  Interventions: Drug: Acetaminophen
- Ibuprofen-acetaminophen combination (Experimental): Ibuprofen 800 mg plus acetaminophen 1 gm
  Interventions: Drug: Ibuprofen-acetaminophen combination

INTERVENTIONS:
Drug: Ibuprofen — single dose
  Other Names: motrin
  Arms: Ibuprofen
Drug: Acetaminophen — single dose
  Other Names: tylenol
  Arms: Acetaminophen
Drug: Ibuprofen-acetaminophen combination — single dose
  Other Names: motrin; tylenol
  Arms: Ibuprofen-acetaminophen combination

SUMMARY:
The purpose of this study is to determine whether the combination of ibuprofen and acetaminophen, is more effective than either single agent alone in treating pain from acute musculoskeletal injuries in the emergency department.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the combination of ibuprofen and acetaminophen, is more effective than either single agent alone in treating pain from acute musculoskeletal injuries in the emergency department. We hypothesize that the combination will be more effective than either agent alone in patients presenting to the emergency department with acute pain from musculoskeletal injuries such as sprain, and bruises. While each agent alone is effective to some degree, many patients do not find complete relief with them and often narcotic agents (with all of their potential side effects) are added. In this study patients experiencing any pain will be randomly given either ibuprofen OR acetaminophen OR their combination and their degree of pain severity will be measured every 15 minutes up to one hour. At the end of this 1 hour patients still experiencing pain and requiring additional pain relief will receive additional analgesics at the discretion of their treating physician. We will not only measure how much the pain severity was reduced but also the percentage of patients that require some form of additional or "rescue" medication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who presented to the emergency department with pain (a verbal numeric pain score greater than 0 on a scale of 0 to 10 from none to greatest) secondary to an acute musculoskeletal injury of less than 24 hours of duration when one of the study investigators was present were eligible for enrollment

Exclusion Criteria:

* Patients who had taken an opioid containing analgesic as well as those with a prior history of allergy or contraindications to ibuprofen or acetaminophen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Singer, MD, Principal Investigator — Stony Brook University

REFERENCES:
- [Derived] Jones P, Lamdin R, Dalziel SR. Oral non-steroidal anti-inflammatory drugs versus other oral analgesic agents for acute soft tissue injury. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007789. doi: 10.1002/14651858.CD007789.pub3. PMID 32797734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the emergency department over a 1 year period
Period: Overall Study
Arm/Group | Ibuprofen | Acetaminophen | Ibuprofen-acetaminophen Combination
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Acetaminophen | Ibuprofen-acetaminophen Combination | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 28 | 86
  >=65 years | 2 | 0 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (16) | 34 (12) | 37 (17) | 36 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 15 | 41
  Male | 16 | 18 | 15 | 49
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: Pain score on 100 mm VAS from 0 (no pain) to 100 (worst pain)
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Ibuprofen | Acetaminophen | Ibuprofen-acetaminophen Combination
Number analyzed (Participants) | 30 | 30 | 30
mm | 39 [28 to 50] | 43 [33 to 53] | 42 [32 to 51]

2. Secondary Outcome: Need for Rescue Pain Relief
Description: The need for additional analgesics
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Ibuprofen | Acetaminophen | Ibuprofen-acetaminophen Combination
Number analyzed (Participants) | 30 | 30 | 30
participants | 11 | 10 | 5

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Ibuprofen | Acetaminophen | Ibuprofen-acetaminophen Combination
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen (N=30) | Acetaminophen (N=30) | Ibuprofen-acetaminophen Combination (N=30)
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Small sample size, single center, short follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No